CLINICAL TRIAL: NCT01490749
Title: Phase I/IIB Study of Induction Chemotherapy With XELOX, Followed by Radiation Therapy and Dose Escalation of RAD001 in Patients With Esophageal Cancer
Brief Title: Trial of XELOX Followed by Radiation Combined With Carboplatin and RAD001 for Esophageal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Nabil F. Saba, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00047026; WCI1871-10 (Other: Other)
Record Dates: First submitted 2011-10-25; First posted 2011-12-13 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Esophageal Cancer; Neoplasms, Esophageal
Keywords: Esophageal Cancer; Neoplasms, Esophageal
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Everolimus; XELOX; Oxaliplatin; Capecitabine; Carboplatin; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- XELOX/Radiation/Carboplatin/RAD001 (Experimental): Patients receive XELOX comprising oxaliplatin intravenously (IV) over 120 minutes on day 1 and capecitabine orally (PO) twice daily (BID) on days 1-14. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo radiotherapy (RT) 5 days a week for up to 6 weeks. Patients also receive carboplatin IV over 15 minutes to 24 hours once weekly for 5-6 weeks and RAD001 PO every other day (QOD) or once daily (QD) for 5-6 weeks during radiation therapy (RT). Patients with resectable disease undergo surgery.
  Interventions: Drug: RAD001; Drug: XELOX; Drug: Carboplatin; Radiation: Radiation

INTERVENTIONS:
Drug: RAD001 — Dose escalation for Phase I; dose for Phase II to be determined after Phase I is completed.
  Other Names: Everolimus
Drug: XELOX — Patients will receive two cycles of XELOX.
  Other Names: Oxaliplatin and capecitabine; Eloxatin and Xeloda
Drug: Carboplatin — Given on a 3 weeks on and 1 week off schedule.
  Other Names: Paraplatin
Radiation: Radiation — 1.8 Gy to 36 Gy; 3 fields or laterals to 50.4 Gy.

SUMMARY:
The purpose of this study is to test the drug RAD001 in combination with another chemotherapy drug, Carboplatin, as well as radiation therapy in the treatment of esophageal cancer. Because RAD001 has not been used in this combination before, it is not clear which dose will be best when used in combination.

The standard of care for patients who have esophageal cancer that has not moved to other areas of the body (non-metastatic) includes a combination of chemotherapy, radiation therapy and possibly surgery. If the patient chooses to participate in this study, the patient will receive chemotherapy and radiation therapy. The patient will possibly also have surgery to have the cancer removed. This decision will be made by the treating physicians. All of the chemotherapy the patient will receive on the study is considered standard chemotherapy for esophagus cancer. The investigators do not know as of yet if the drug called RAD001 will help improve the treatment for patients with this disease. RAD001 is a pill that has been used in many other types of cancer and has been proven to be effective in other cancers such as kidney cancer.

DETAILED DESCRIPTION:
Esophageal cancer is the sixth most common cause of cancer-related death worldwide. Recent medical advances have led to small improvements in survival, but the overall rate of survival remains low, making new treatment approaches necessary.

Chemotherapy drugs and radiation therapy are often both used in treating esophageal cancer. The combination of oxaliplatin and capecitabine (XELOX) is a commonly used chemotherapy combination. Sometimes chemotherapy is given as an "induction" therapy, before the radiation is given.

The drug RAD001 is a targeted drug that acts specifically on a protein inside cells (called mTOR), which is important for cancer development. The combination of RAD001 and radiation therapy has been shown to improve anti-cancer effects.

This study will look for the ideal dose of RAD001 when given in combination with radiation therapy after induction chemotherapy with XELOX, and test the anticancer effects of this treatment approach in patients with esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed squamous cell carcinoma or adenocarcinoma of the esophagus or gastroesophageal (GE) junction.
* Patients can have disease that is resectable or unresectable.
* Patients must not have had prior chemotherapy or radiation therapy for esophageal cancer.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Age ≥ 18.
* Adequate bone marrow, liver and renal function as assessed by the following:

  * Absolute neutrophil count (ANC) ≥ 1500/mm³.
  * Platelet count ≥ 100,000/mm³.
  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN).
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN (≤ 5 x ULN for patients with liver involvement).
  * Creatinine ≤ 1.5 x ULN.
* Fasting serum cholesterol ≤ 300 mg/dL OR ≤ 7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
* Women of childbearing potential must have a negative pregnancy test prior to first receiving investigational product. Sexually active women of childbearing potential (WOCBP) must use an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized. All WOCBP should be instructed to contact the Investigator immediately if they suspect they might be pregnant (e.g., missed or late menstrual period) at any time during study participation.
* Patient must be willing to sign informed consent.

Exclusion Criteria:

* Patients currently receiving other investigational agents.
* Patients with known distant metastases.
* Patients who have received prior treatment with an mammalian target of rapamycin (mTOR) inhibitor (sirolimus, temsirolimus, everolimus).
* Patients with a known hypersensitivity to RAD001 (everolimus) or other rapamycins (sirolimus, temsirolimus) or to its excipients.
* Known hypersensitivity to oxaliplatin, other platinum-containing compounds.
* Patients with known brain metastases.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as a known history of HIV seropositivity.
* History of active hepatitis B or C.
* Co-administration with strong inhibitors of cytochrome P450 3A4 isoenzyme (CYP3A4) (e.g., ketoconazole, itraconazole, ritonavir) or P-glycoprotein (PgP).
* Patients with an active, bleeding diathesis.
* Patients with significant intercurrent medical illness (including New York Heart Association [NYHA] class III or IV heart disease, significant arrhythmias requiring medication, symptomatic coronary artery disease, myocardial infarction) within the previous 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Phase I portion to determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of RAD001 in combination with radiation | within one month after surgery

SECONDARY OUTCOMES:
Rate of surgical pathologic complete remission (pCR) (absence of evidence of cancer after surgery) | within one month from surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nabil F. Saba, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (3):
- United States (3):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Vanderbilt University, Nashville, Tennessee